CLINICAL TRIAL: NCT03309644
Title: Comparative Effectiveness of Peripheral Nerve Blocks for Outpatient Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GMH1
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Complications
Keywords: Unplanned admissions; Visits to the ED; Readmissions; Death
MeSH Terms: conditions — Postoperative Complications; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripheral nerve block: Peripheral nerve block
  Interventions: Other: Peripheral nerve blockade
- No peripheral nerve block: No peripheral nerve block
  Interventions: Other: No peripheral nerve blockade

INTERVENTIONS:
Other: Peripheral nerve blockade — Participants who receive a peripheral nerve block identified through the medical chart.
  Groups: Peripheral nerve block
Other: No peripheral nerve blockade — Participants who did not receive a peripheral nerve block identified through the medical chart.
  Groups: No peripheral nerve block

SUMMARY:
This retrospective, population-based cohort study will evaluate the comparative effectiveness of peripheral nerve blocks on patient outcomes after ambulatory shoulder surgery in adults patients undergoing surgery in Ottawa, Ontario.

DETAILED DESCRIPTION:
The investigators will use a coarsened exact matching algorithm prior to the analysis to minimize bias in this observational study. A multivariate logistic regression model will be used to compare the effect of anesthesia interventions on the primary outcome within matched cohorts. Sensitivity analyses will be used to evaluate the robustness of the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Ontario residents
* Aged 18 years and older
* Elective ambulatory shoulder surgery

Exclusion Criteria:

* Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective, population-based, cohort study based in Ottawa, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 1623 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I McIsaac, MD, MPH, Principal Investigator — Department of Anesthesiology and Pain Medicine, University of Ottawa
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton GM, Ramlogan R, Lui A, McCartney CJL, Abdallah F, McIsaac DI. Association of peripheral nerve blocks with postoperative outcomes in ambulatory shoulder surgery patients: a single-centre matched-cohort study. Can J Anaesth. 2019 Jan;66(1):63-74. doi: 10.1007/s12630-018-1234-8. Epub 2018 Oct 17. PMID 30334192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Nerve Block | No Peripheral Nerve Block
Started | 1382 | 241
Completed | 1382 | 241
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Block | No Peripheral Nerve Block | Total
Number analyzed (Participants) | 1382 | 241 | 1623
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (15.4) | 47.1 (15.4) | 49.7 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455 | 86 | 541
  Male | 927 | 155 | 1082
Year of Surgery [Count of Participants; unit: Participants]
  2011/12 | 517 | 131 | 648
  2013/14 | 422 | 74 | 496
  2015/16 | 443 | 36 | 479
Elixhauser comorbidity index [Count of Participants; unit: Participants] — The Elixhauser Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases diagnosis codes. Each comorbidity category is documented as disease presence or disease absence and there are 31 categories. Therefore, a higher score indicates more presence of disease (with 31 being the maximum).
  Participants
    < 0 | 0 | 0 | 0
    0 | 1380 | 240 | 1620
    1-5 | 0 | 0 | 0
    > 5 | 0 | 0 | 0
    Unable to report due to small cell size | 2 | 1 | 3
Surgery Location [Count of Participants; unit: Participants]
  Shoulder joint | 852 | 188 | 1040
  Rotator cuff | 528 | 45 | 573
  Shoulder muscle | 2 | 8 | 10
American Society of Anesthesiology (ASA) Score [Count of Participants; unit: Participants] — Physical status classification used to determine a patient's risk with anaesthesia. The score ranges from I to VI, with I indicating a healthy person and VI indicating a deceased organ donor. A higher score indicates greater risk. Population: Six missing values for ASA score, all from the 'No PNB' group
  Participants
    < 2: number analyzed (Participants) | 1382 | 235 | 1617
    < 2 | 1054 | 183 | 1237
    > 2: number analyzed (Participants) | 1382 | 235 | 1617
    > 2 | 328 | 52 | 380
Surgery type [Count of Participants; unit: Participants]
  Arthroscopic | 1297 | 212 | 1509
  Open | 85 | 29 | 114
Campus [Count of Participants; unit: Participants]
  Civic | 143 | 24 | 167
  General | 487 | 129 | 616
  Riverside | 752 | 88 | 840

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complication
Description: Composite outcome: 1) unplanned admissions on the day of surgery, 2) post-discharge ED visits within 30 days of surgery, 3) readmission within 30 days of surgery, and 4) death from any cause.
Time Frame: From day of surgery to 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block | No Peripheral Nerve Block
Number analyzed (Participants) | 1382 | 241
Participants
  Composite outcome | 130 | 23
  Unplanned admission | 20 | 12
  Readmission within 30 days | 11 | 3
  ED visits within 30 days | 111 | 11

2. Secondary Outcome: Health System Costs in the 30 Days After Surgery
Description: Calculated using validated algorithms
Time Frame: From day of surgery to 30 days after surgery
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Peripheral Nerve Block | No Peripheral Nerve Block
Number analyzed (Participants) | 1357 | 231
dollars | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality was collected including all deaths both anticipated and unanticipated due to any cause. Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Peripheral Nerve Block | No Peripheral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/1382 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There is risk of exposure misclassification bias. Confounding bias may have influenced the receipt of specific anesthesia interventions and outcomes. This study did not examine longer-term outcomes. We do not have data that specifically link the anesthesiologist or surgeon to the patient. This study examines data obtained from a single academic health sciences centre. Given the unexpected lower rates of adverse events in our institution, results may be due to this study being underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No